CLINICAL TRIAL: NCT07222423
Title: Epidemiology and Hospital Management of Patients With PROS in France: a PMSI Study
Brief Title: A Study of the Epidemiology and Hospital Management of Patients With PROS in France
Acronym: EpiPROS
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBYL719F1FR02
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: PIK3CA-Related Overgrowth Spectrum
Keywords: PIK3CA; Prevalence; Healthcare Resource Consumption; Cost
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Target Population (P1): Children and adults hospitalized for disease management of PROS.
- Subpopulation (SP1): Patients from P1 with at least two PROS-related hospitalizations (including the index hospitalization).

SUMMARY:
The purpose of this study was to estimate the incidence and prevalence of a group of genetic disorders known as PIK3CA-Related Overgrowth Spectrum (PROS) in France. Additionally, the study aimed to characterize patients, disease management, and costs associated with PROS. This study used data from the French National Hospitals Database, Programme de Médicalisation des Systèmes d'Information (PMSI). The study period was from January 2015 to December 2022.

ELIGIBILITY:
Inclusion criteria:

Population P1 was identified using a combined query, considering:

* International Classification of Diseases, 10th Revision, Clinical Modification (ICD-10-CM) codes for PROS-related malformations; OR
* PROS-related technical procedures performed during hospitalizations to relieve the symptoms of the disease.

Subpopulation SP1 was identified through the identification of at least two PROS-related hospitalizations (PROS-related ICD-10-CM or technical procedure code), including the index hospitalization.

Exclusion criteria:

Presence at any time during the entire study period of:

* ICD-10-CM codes for chromosomal malformation; OR
* ICD-10-CM code for hemangioma to avoid inclusion of patients with hemangioma and other vascular malformation; OR
* ICD-10-CM codes associated with the following comorbidities: cancer, cerebrovascular pathologies, hemiplegia (for pediatric patients only), metastatic pathologies, or myocardial infarction.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 3605 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Yearly Prevalence Rate | Up to approximately 6 years
  Yearly prevalence rate was calculated by dividing the number of identified patients with PROS by the total French population during the inclusion period. The inclusion period was from January 2017 to December 2022.
Yearly Incidence Rate | Up to approximately 6 years
  Yearly incidence rate was calculated by dividing the number of PROS newly diagnosed cases during the inclusion period (incident cases) by the total French population during the inclusion period. The inclusion period was from January 2017 to December 2022.

SECONDARY OUTCOMES:
Number of Patients by Patient Characteristics | Baseline
  Patient characteristics included age, sex, region of residence, and comorbidities.
Number of Comorbidities per Patient | Baseline
Number of Patients by PROS Diagnosis | Baseline
  Diagnoses included:
  * Lymphangioma, any site
  * Peripheral arteriovenous malformation
  * Arteriovenous malformation of precerebral vessels
  * Arteriovenous malformation of the cerebral vessels
  * Megalencephaly
  * Other congenital malformations of the upper limb(s), including the shoulder girdle [Macrodactyly (fingers)]
Number of Patients by Type of PROS-related Technical Procedures | Baseline
  Technical procedures were identified by codes according to the Medical Classification for Clinical Procedure Nomenclature (CCAM).
Number of Patients by Type of Hospitalization | Baseline
  Hospitalization type included inpatient and outpatient visits.
Average Length of Stay of Hospitalization | Baseline
Number of Patients by Hospitalization Severity | Baseline
  The severity of a hospitalization was determined by the values 1/2/3/4 assigned to the last character of the Diagnosis Related Group (DRG) code for that hospitalization, with higher numbers indicating greater severity.
Average Duration of Follow-up | Up to approximately 6 years
Number of All-cause Hospitalizations During the Follow-up Period | Up to approximately 6 years
  All-cause hospitalizations included medical, surgery, obstetrics and dentistry.
Number of PROS-related Hospitalizations During the Follow-up Period | Up to approximately 6 years
  PROS-related hospitalizations included outpatient and inpatient hospitalizations.
Average Length of Stay of PROS-related Inpatient Hospitalization During the Follow-up Period | Up to approximately 6 years
Number of Patients With PROS-related Hospitalization During the Follow-up Period by Type of Hospitalization and Age Range | Up to approximately 6 years
  Hospitalizations included inpatient and outpatient hospitalizations.
Number of PROS-related Hospitalizations by Year of Follow-up | Up to approximately 6 years
Number of PROS-related Hospitalizations During the Follow-up Period by Level of Severity | Up to approximately 6 years
  The severity of a hospitalization was determined by the values 1/2/3/4 assigned to the last character of the DRG code for that hospitalization, with higher numbers indicating greater severity.
Number of All-cause External Technical Procedures and Visits During the Follow-up Period | Up to approximately 6 years
Number of Patients With at Least one All-cause External Technical Procedure and Visit During the Follow-up Period | Up to approximately 6 years
Number of External Technical Procedures and Visits of Interest During the Follow-up Period | Up to approximately 6 years
  Procedures and visits of interest were under the following specialties:
  * Psychiatry
  * Dental surgery
  * Vascular medicine
  * Medical genetics
  * Hematology
  * Nephrology
  * Visceral and digestive surgery
  * Gastroenterology and hepatology
  * Reconstructive and aesthetic plastic surgery
  * Orthopedic surgery and traumatology
  * Pediatric surgery
  * Dermatology and venereology
  * Pediatrics
  * Anesthesiology
  * Nurse
  * Radiodiagnostic and medical imaging
Number of Patients With an External Technical Procedure and Visit of Interest During the Follow-up Period | Up to approximately 6 years
  Procedures and visits of interest were under the following specialties:
  * Psychiatry
  * Dental surgery
  * Vascular medicine
  * Medical genetics
  * Hematology
  * Nephrology
  * Visceral and digestive surgery
  * Gastroenterology and hepatology
  * Reconstructive and aesthetic plastic surgery
  * Orthopedic surgery and traumatology
  * Pediatric surgery
  * Dermatology and venereology
  * Pediatrics
  * Anesthesiology
  * Nurse
  * Radiodiagnostic and medical imaging
Number of External Technical Procedures and Visits by Specialty of the Performing Healthcare Professional During the Follow-up Period | Up to approximately 6 years
  Healthcare professional specialties included:
  * Psychiatry
  * Dental surgery
  * Vascular medicine
  * Medical genetics
  * Hematology
  * Nephrology
  * Visceral and digestive surgery
  * Gastroenterology and hepatology
  * Plastic, reconstructive, and aesthetic surgery
  * Orthopedic surgery and traumatology
  * Pediatric surgery
  * Dermatology and venereology
  * Pediatrics
  * Anesthesiology
  * Nurse
  * Radiodiagnostic and medical imaging
Number of Emergency Room Visits not Followed by Hospitalization During the Follow-up Period | Up to approximately 6 years
Number of Patients With at Least one Emergency Room Visit not Followed by Hospitalization During the Follow-up Period | Up to approximately 6 years
Healthcare Resource Consumption Rate Per Patient-Year (PPY) During the Follow-up Period | Up to approximately 6 years
  Healthcare resource consumption rates PPY were calculated by dividing the sum of the number of hospital care visits for the patients of interest by the sum of the years of follow-up for all these patients. Rates were calculated for:
  * All-cause hospitalization
  * PROS-related hospitalization (inpatient and outpatient)
  * All-cause external technical procedures and visits
  * External technical procedures and visits performed by healthcare professionals of interest
  * Emergency room visits not followed by hospitalization
Healthcare Costs PPY During the Follow-up Period | Up to approximately 6 years
  Healthcare costs PPY were calculated by dividing the sum of the hospital costs for the patients of interest by the sum of the years of follow-up for all these patients. Costs were calculated for:
  * All-cause hospitalization
  * All-cause external technical procedures and visits
  * PROS-related hospitalization
  * External technical procedures and visits performed by healthcare professionals of interest

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States